CLINICAL TRIAL: NCT01960738
Title: A Group Randomized Trial to Evaluate the Efficacy of Using Pre-dive Checklist to Prevent the Incidence of Recreational Scuba Diving Mishaps
Brief Title: Common Recreational Diving Practices: A Randomized Control Trial Using Pre-Dive Checklist
Acronym: Checklists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Divers Alert Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DAN009-12
Record Dates: First submitted 2013-10-07; First posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Injuries
Keywords: Diving; Water; Recreation; Precursor
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Intervention (Experimental): The intervention group received a pre-dive checklist and a post-dive log
  Interventions: Other: A pre-dive checklist
- Control (No Intervention): The control group received the post-dive log only.

INTERVENTIONS:
Other: A pre-dive checklist — The pre-dive checklist included a checklist of tasks to be undertaken before the dive, a dive-plan that asked the diver to plan the depth, and amount of gas kept at different levels of diving, and 4 dive tips.
  Arms: Intervention

SUMMARY:
To evaluate the efficacy of using a pre-dive checklist to prevent the incidence of diving mishaps in recreational divers.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Having a valid Diver Certification
* Deemed fit by the Dive operator to dive on the day of participation
* Planning to dive on the day of participation
* Have basic knowledge of English

Exclusion Criteria:

* Anyone not meeting all of the inclusion criteria
* A diver who did not answer the outcomes questionnaire was later excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Mishaps | One day
  Mishaps were reported by scuba divers themselves, at the end of their diving day (the day they were enrolled). Mishaps are precursors of injuries. Injuries are less common outcomes (in fact, nobody got injured), hence we used mishaps - which allowed us to test the efficacy of pre-dive checklists, and do so with limited resources.

SECONDARY OUTCOMES:
Major mishaps | One day
  Major mishaps are a type of mishaps
Minor Mishaps | One day
  Minor mishaps are a type of mishaps

CONTACTS AND LOCATIONS:
Overall Officials: Shabbar I Ranapurwala, MPH, Principal Investigator — Research Assistant, Medical Research; Petar J Denoble, MD, DSc, Study Director — Vice President, Medical Research
Locations (4):
- Aquatic Safaris, Wilmington, North Carolina, United States
- Sunset House, George Town, Grand Cayman, Cayman Islands
- Mexico (2):
  - Aldora Divers, San Miguel de Cozumel, Quintana Roo
  - Sand Dollar Sports, San Miguel de Cozumel, Quintana Roo

REFERENCES:
- [Derived] Ranapurwala SI, Denoble PJ, Poole C, Kucera KL, Marshall SW, Wing S. The effect of using a pre-dive checklist on the incidence of diving mishaps in recreational scuba diving: a cluster-randomized trial. Int J Epidemiol. 2016 Feb;45(1):223-31. doi: 10.1093/ije/dyv292. PMID 26534948